CLINICAL TRIAL: NCT04956718
Title: Breath Metabolomics of Placebo Effects Via Cold Pressor Test
Brief Title: Breath Metabolomics of Placebo Effects, a Pilot Study
Acronym: BMPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-01132; ks21Sinues
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Analgesia
Keywords: pain; placebo effects; analgesia; placebo analgesia; cold pressor test; breath metabolomics
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Intervention Model Description: Single centered; national ,randomized, crossover, pilot study
Who Masked: Participant
Masking Description: participants do not know its a placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPT first (Other): Cold Pressor Test (CPT): apparatus for the task is a tank of water of temperature of 4 °C (+-0.5 °C), with instruction to immerse the hand until too uncomfortable to continue. A maximum time limit per immersion of 3-5 min is applied. Quantitative measurement can then be made of pain threshold (point first perceived as painful) and tolerance time.
  All 20 participants will undergo two study visits. The order in which they will receive CPT and CPT plus placebo differs, with participants being randomly split into two groups. 10 participants first CPT + placebo and then CPT, and 10 participants vice versa.
  Interventions: Other: Cold Pressor Test (CPT); Other: Placebo NaCl Nasal spray
- CPT+placebo first (Other): Participant will be told and read about the 'pain medication' (= Placebo NaCl Nasal spray). Thereafter participant will self-administer a nasal spray, which is in fact a placebo nasal spray containing NaCl solution and Cold Pressor Test (CPT) is performed.
  All 20 participants will undergo two study visits. The order in which they will receive CPT and CPT plus placebo differs, with participants being randomly split into two groups. 10 participants first CPT + placebo and then CPT, and 10 participants vice versa
  Interventions: Other: Cold Pressor Test (CPT); Other: Placebo NaCl Nasal spray

INTERVENTIONS:
Other: Cold Pressor Test (CPT) — Cold Pressor Test (CPT): apparatus for the task is a tank of water of temperature of 4 °C (+-0.5 °C), with instruction to immerse the hand until too uncomfortable to continue. A maximum time limit per immersion of 3-5 min is applied. Quantitative measurement can then be made of pain threshold (point first perceived as painful) and tolerance time.
Other: Placebo NaCl Nasal spray — placebo nasal spray containing NaCl solution

SUMMARY:
This study is to analyze the breath metabolome before and after the administration of a placebo in an established experimental pain procedure in healthy subjects in order to investigate placebo effects, and whether they induce any measurable changes at the metabolic level.

DETAILED DESCRIPTION:
Interrogation of the exhaled breath metabolome will be performed by using an objective method of measurement for placebo effects in pain analgesia, known as Cold Pressure Test (CPT). CPT reactions can be measured objectively by blood pressure spikes as well as changes in continuous heart rate monitoring.To this end, probands will be continuously connected to a Heartrate & Blood Pressure Monitor. First, baseline exhalation will be assessed. Then, the CPT is performed according to the 'CPT Guide' with subsequent post-pain exhalations analysis with or without self-administration of the placebo (NaCl nasal spray). After 15 minutes rest, probands will be submitted to a second post-pain exhalations set (+/- placebo). The process is completely non-invasive as the participant just exhales through a commercially available disposable bacterial/viral filter coupled to the ion source.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male adult volunteers
* German speaking, or good knowledge of the German language
* Able to understand the study
* Able to give informed consent

Exclusion criteria:

* Regularly taking medication potentially interfering with pain sensation (analgesics, antihistamines and calcium and potassium channel blockers)
* Current pregnancy
* Daily smokers (as per WHO definition: A daily smoker is someone who smokes any tobacco product at least once a day.)
* Neuropathy
* Chronic pain
* Neuromuscular or psychiatric disease
* Known or suspected heart, kidney or liver disease
* Hypertension (Systolic (mmHg) >130, Diastolic (mmHg) >80)
* History of fainting or seizures
* History of Frostbite
* Current medications (psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
change in signal intensity of mass-to-charge ratio (m/z) of exhaled metabolites | 1 hour
  The variable of primary interest is the variation of signal intensity of mass-to-charge ratio (m/z) of exhaled metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sinues, Prof. Dr., Principal Investigator — Universitäts-Kinderspital beider Basel (UKBB)
Locations (1):
- Universitäts-Kinderspital beider Basel (UKBB), Basel, Canton of Basel-City, Switzerland